CLINICAL TRIAL: NCT07242469
Title: A Multiple Dose Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of MK-1403 in Participants With Type 2 Diabetes Mellitus
Brief Title: A Clinical Trial of MK-1403 in Participants With Type 2 Diabetes Mellitus (MK-1403-006)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 1403-006
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Panel A MK-1403 + additive coformulation dose 1 (Experimental): Participants will receive MK-1403 + additive coformulation dose 1 orally once daily.
  Interventions: Drug: MK-1403 + additive coformulation
- Panel A Placebo + additive coformulation dose 1 (Placebo Comparator): Participants will receive Placebo + additive coformulation dose 1 orally once daily.
  Interventions: Drug: Placebo + additive coformulation
- Panel B MK-1403 + additive coformulation dose 2 (Experimental): Participants will receive MK-1403 + additive coformulation dose 2 orally once daily
  Interventions: Drug: MK-1403 + additive coformulation
- Panel B Placebo + additive coformulation dose 2 (Placebo Comparator): Participants will receive Placebo + additive coformulation dose 2 orally once daily
  Interventions: Drug: Placebo + additive coformulation

INTERVENTIONS:
Drug: MK-1403 + additive coformulation — MK-1403 + additive coformulation is a co-formulated product of MK-1403 administered orally.
  Arms: Panel A MK-1403 + additive coformulation dose 1; Panel B MK-1403 + additive coformulation dose 2
Drug: Placebo + additive coformulation — Placebo + additive coformulation is a co-formulated product of placebo administered orally.
  Arms: Panel A Placebo + additive coformulation dose 1; Panel B Placebo + additive coformulation dose 2

SUMMARY:
The purpose of this study is to learn about the safety and if people tolerate a study medicine called MK-1403. The study will also measure what happens to MK-1403 in the body of a person with type 2 diabetes (T2D) over time (pharmacokinetic or PK study), and how it affects the amount of high-sensitivity C-reactive protein (hsCRP) in a person's blood.

ELIGIBILITY:
Inclusion Criteria:

* Has a confirmed diagnosis of Type 2 diabetes mellitus (T2DM)
* Has body mass index (BMI) between 18 and 40 kg/m^2, inclusive

Exclusion Criteria:

* Has Type 1 diabetes mellitus or secondary types of diabetes
* Has a history of congestive heart failure (New York Heart Association [NYHA] Class 3 or 4)
* Has history of myocardial infarction, uncontrolled arrhythmias, cardiac revascularization, angina, unstable peripheral arterial disease and/or stroke
* Has history of cancer (malignancy)
* Has positive test(s) for hepatitis B surface antigen (HBsAg), hepatitis C antibodies, or human immunodeficiency virus (HIV)
* Has a history of gastrointestinal (GI) disease which might affect food and drug absorption, or has had gastric bypass or similar surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-12-22 (Actual); Primary Completion 2026-08-28 (Estimated); Study Completion 2026-08-28 (Estimated)

PRIMARY OUTCOMES:
Number of participants who experience one or more adverse events (AE) | Up to approximately 28 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience one or more AEs will be reported.
Number of participants who discontinue study intervention due to adverse events | Up to approximately 14 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study intervention due to an AE will be reported.

SECONDARY OUTCOMES:
Change from Baseline in Placebo-Corrected High Sensitivity C-Reactive Protein (hsCRP) Serum Concentration | Baseline and 24-hours postdose on Day 14
  Blood samples will be collected to determine the change from baseline in placebo-corrected hsCRP.
Plasma concentration of MK-1403 at 24 Hours Postdose (C24) on Day 14 | 24-hour postdose on Day 14
  Blood samples will be collected to determine the C24 of MK-1403 in plasma on Day 14.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (4):
- United States (4):
  - ProSciento Inc. ( Site 0001), Chula Vista, California
  - QPS-MRA, LLC ( Site 0004), Miami, Florida
  - Advanced Pharma CR, LLC ( Site 0003), Miami, Florida
  - Bio-Kinetic Clinical Applications, LLC dba QPS-MO ( Site 0005), Springfield, Missouri

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com